CLINICAL TRIAL: NCT04456309
Title: Brain MRI Characteristics in Stroke Patients With Intracardiac Thrombus
Brief Title: Brain MRI in Stroke Patients With Intracardiac Thrombus
Acronym: BRAIN IRM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2020/DR-02
Record Dates: First submitted 2020-06-22; First posted 2020-07-02 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Intracardiac Thrombus
Keywords: brain MRI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atrial fibrillation: stroke patients with atrial fibrillation
  Interventions: Other: No intervention,
- Intracardiac thrombus: stroke patients with intracardiac thrombus
  Interventions: Other: No intervention,

INTERVENTIONS:
Other: No intervention, — pure observational study

SUMMARY:
Acute infarction patterns have been described in cardioembolic stroke, mainly with atrial fibrillation (AF) or patent foramen ovale. We aimed to analyse acute infarction MRI characteristics in stroke patients with intracardiac thrombus (ICT) compared with stroke patients with AF.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients presenting with acute symptomatic cardioembolic infarction associated with ICT, recruited and registered in the stroke database between June 2018 and November 2019 of our centre (Nîmes University Hospital, France). These patients were compared with consecutive cardioembolic stroke patients with known or newly discovered AF (in the absence of ICT on echocardiography), recruited during the same time period.
* Brain MRI (including diffusion-weighted imaging [DWI]) performed within one week of symptom onset; complete etiological work-up including intracranial (time-of-flight [TOF], gadolinium-enhanced magnetic resonance angiography [MRA], or computed tomographic angiography [CTA]) and extracranial (gadolinium-enhanced MRA, CTA, or duplex ultrasound) vessel imaging; transthoracic or transoesophageal echocardiography; and ≥24h ECG monitoring (acute stroke unit monitoring and/or Holter ECG monitoring).

Exclusion Criteria:

* opt-out patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 groups of patients :
  1 - Stroke patients with atrial fibrillation
  2- Stroke patients with intracardiac thrombus
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Brain MRI characteristics | Day of inclusion (Day 1)
  infarction location (anterior/middle/posterior cerebral artery territory; anterior/posterior/mixed anterior-posterior circulation; multiterritorial infarction; brainstem; cerebellum; small cortical cerebellar infarctions [SCCI] or non-SCCI; cortical/subcortical/corticosubcortical)
Brain MRI characteristics | Day of inclusion (Day 1)
  lesion number
Brain MRI characteristics | Day of inclusion (Day 1)
  subcortical lesion size (><15 mm)
Brain MRI characteristics | Day of inclusion (Day 1)
  total infarction volume.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri RENARD, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Renard D, Castelnovo G, Ion I, Guillamo JS, Thouvenot E. Single and simultaneous multiple intracerebral hemorrhages: a radiological review. Acta Neurol Belg. 2020 Aug;120(4):819-829. doi: 10.1007/s13760-020-01385-4. Epub 2020 May 24. PMID 32449137
- [Derived] Trandafir C, Sandiramourty S, Laurent-Chabalier S, Ter Schiphorst A, Nguyen H, Wacongne A, Ricci JE, Pereira F, Thouvenot E, Renard D. Brain Infarction MRI Pattern in Stroke Patients with Intracardiac Thrombus. Cerebrovasc Dis. 2021;50(5):581-587. doi: 10.1159/000515707. Epub 2021 Jun 17. PMID 34139688